CLINICAL TRIAL: NCT05915455
Title: Face and Content Validation of a Healthcare Professional-facing Toolkit to Communicate Information on the Portfolio Diet and PortfolioDiet.app
Brief Title: HCP-facing Portfolio Diet Toolkit Validation Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Laura Chiavaroli, Prinicipal Investigator, University of Toronto
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HCPTestPD2023
Record Dates: First submitted 2023-06-09; First posted 2023-06-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Cardiovascular Diseases
Keywords: Portfolio Diet; Cardiovascular Disease; Risk Reduction
MeSH Terms: conditions — Cardiovascular Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- HCP resource evaluation (Experimental): HCP will be provided with resources to evaluate
  Interventions: Other: HCP-facing Portfolio Diet Infographic + Informative Video; Other: Portfolio Diet Application

INTERVENTIONS:
Other: HCP-facing Portfolio Diet Infographic + Informative Video — Resources to evaluate include the healthcare professional-facing Portfolio Diet infographic (1-page) and 4-minute accompanying video
Other: Portfolio Diet Application — Resource to evaluate includes the Portfolio Diet mobile application

SUMMARY:
There is limited support in primary care for diet and lifestyle, the cornerstones for therapy in clinical practice guidelines. Canadian dietitian services are not covered by provincial health plans and most physicians cite a lack of education, tools and time to counsel on nutrition. To engage healthcare professionals (HCP) and patients in the delivery of nutrition interventions, the investigators have developed the Portfolio Diet mobile application, as a direct translation of clinical practice guidelines for cardiovascular and diabetes risk reduction which recommend the Portfolio Diet, a plant-based dietary pattern of cholesterol-lowering foods. To increase confidence and comfortability in advising patients on the Portfolio Diet, the investigators have developed an HCP-facing toolkit (infographic and video) to communicate information on the Portfolio Diet and Portfolio Diet mobile application. To ensure validity of these resources, the investigators will conduct face and content validation of the HCP-facing toolkit and assess whether it increases HCP knowledge and potential use in practice, and assess HCP perspectives on the Portfolio Diet mobile application.

DETAILED DESCRIPTION:
Background:

As the Canadian population ages, there is an increased risk of cardiovascular disease (CVD) and higher healthcare costs. Thus, there is a need for dietary approaches to target these challenges. Furthermore, with the transition to greater virtual care, innovative technology-based interventions using mobile applications provide an opportunity to engage healthcare professionals (HCP), including family physicians, registered dietitians (RDs), nurses, pharmacists, and patients in delivering nutrition care to save time, provide education, and reduce costs. The Portfolio Diet, an evidence-based therapeutic dietary pattern for CVD risk reduction, is uniquely positioned to test this innovative paradigm. This plant-based dietary pattern of five cholesterol-lowering foods (nuts, legumes, viscous fibre, plant sterols, monounsaturated fat) has been shown to result in the same low-density lipoprotein-cholesterol (LDL-C) and C-reactive protein reductions (CRP) (~30%) as statin therapy in a head-to-head randomized controlled trial. A recent systematic review and meta-analysis. confirmed these effects and showed benefits on other cardiovascular risk factors including non-high-density lipoprotein-cholesterol (non-HDL-C), apoB, triglycerides, and blood pressure. Prospective cohort studies have also shown that the Portfolio Diet is associated with a lower risk of CVD, particularly coronary heart disease, and type 2 diabetes. These benefits have led to widespread recognition of the Portfolio Diet from major international clinical practice guidelines, including the Canadian Cardiovascular Society (CCS). The investigators recently developed the Portfolio Diet mobile application, as a transformative digitally-enabled health service tool for the translation of current CCS guidelines to manage dyslipidemia and prevent CVD.

While the Portfolio Diet is recognized by clinical practice guidelines as a preventive nutrition therapy for CVD, many HCPs remain unaware of the Portfolio Diet and of the Portfolio Diet mobile application. To increase confidence and comfortability in advising patients on the Portfolio Diet, the investigators developed an HCP-facing toolkit (infographic and video) to communicate information on the Portfolio diet and Portfolio Diet app. To ensure validity, the investigators plan to conduct face and content validation of the HCP-facing toolkit and assess whether it increases HCP knowledge and potential use in practice, as well as to assess HCP perspectives of the Portfolio Diet app.

Objectives:

The primary objective is to face and content validate the HCP-facing toolkit and assess whether it increases HCP knowledge and potential use in practice. The second objective is to conduct a quality improvement assessment of the Portfolio Diet mobile application to evaluate its usability, acceptability, knowledge acquisition, quality, and potential use in practice.

Design: We aim to recruit 65 physicians, registered dietitians, and other allied HCP from clinics for a 2-phase study to assess face and content validation of the HCP-facing toolkit and usability of the Portfolio Diet mobile application. In phase 1, 15 HCP with receive the toolkit and a feedback questionnaire. In phase 2, 10 HCPs from phase 1 will be invited to create an account on the Portfolio Diet mobile application and use it daily for 5-minutes over 7-days. On Day 8, a mixed-form questionnaire will be used to evaluate acceptability, knowledge acquisition, engagement, usability using the System Usability Scale (SUS) and the mHealth App Usability Questionnaire (MAUQ), and potential use in practice. After the first round, data will be compiled and reviewed to assess if revisions should be made. Based on the results from the first round, either the original or the revised versions will be presented in the second round to 50 HCP following a similar assessment method as per round 1 but in addition to the SUS and MAUQ, the mixed-form questionnaire will include the Mobile Application Rating Scale (MARS) to assess the quality of the app. This sample size in round 2 was selected to enhance external validity and ensure a representative sample of HCPs, aiding in the validation of the MARS.

Outcomes: The primary outcomes are face and content validation of the HCP-facing toolkit resources. The secondary outcomes are usability, acceptability, knowledge acquisition, engagement, potential use in practice, and the quality of the Portfolio Diet app.

Data analyses: The Phase I feedback questionnaire for the HCP-facing Portfolio diet infographic and video consists of part A to assess content validity of the infographic and parts B and C to assess face validity of the infographic and video, respectively. In part A, the infographic has been divided into 6 parts, which HCP will be asked to rate individually on a scale of one to four with regard to its relevance. In parts B and C, HCP will be asked to rate a series of statements assessing content validity on a scale of 1-5, with 1 being "strongly disagree" and 5 being "strongly agree" for the infographic and video, respectively. After the first round, data will be compiled and reviewed with the study team. Lynn's method will be used to assess content validity of the HCP-facing infographic and video. If more than 30% of respondents rate any question in part A as irrelevant or rate 1-2 for any question in parts B or C, revisions will be made to the HCP-facing Portfolio diet toolkit resources as applicable. The second round of HCP will be presented either the original version or, if >30% rate the resources poorly, the revised version of the toolkit resources will be used and the HCP asked to follow the same method of assessing face and content validity.

In Phase 2, after 7-days of using the Portfolio Diet app, a mixed-form questionnaire will be used to evaluate the acceptability, knowledge acquisition, engagement with the app, usability using the SUS and the MAUQ, and potential use in practice. The SUS is a validated usability questionnaire used in clinical settings to assess the usability of various systems and tools. The SUS includes 10 statements on a 5-point Likert scale, which is a psychometric scale frequently applied in health, and nutrition research, as well as in quality improvement testing, to assess the acceptability of systems and tools. The MAUQ is a recently developed questionnaire that focuses specifically on the usability of mobile health apps. It offers four versions catering to different app types (interactive or standalone) and target app users (patient or HCP), with the HCP-facing versions not yet validated. As such, data will be collected on the standalone HCP-facing version of the MAUQ in addition to the widely used SUS to contribute to validation. The SUS includes 10 statements rated on a 5-point Likert scale. The standalone, HCP-facing MAUQ includes 18 statements rated on a 7-point Likert scale. After the first round, data will be compiled and reviewed with the study team. If the calculated SUS is <70 or more than 30% of respondents indicate serious concerns, revisions will be made to the Portfolio Diet app. The second round of HCP will be presented either the original version or if >30% rate the Portfolio Diet app poorly, the revised version of the Portfolio Diet app to review following the same assessment method with the addition of assessing the quality of the Portfolio Diet app using the MARS. The MARS is a widely used tool for assessing the quality of mobile health apps. It comprises a 19-item objective evaluation across four domains: engagement, functionality, aesthetics, and information. It also includes a 4-item subjective quality assessment, and a specific 6-item section tailored to the app being evaluated, all of which are rated on a 5-point Likert scale specific to each statement.

Hypothesis:

Validating the HCP-facing toolkit will demonstrate support for HCP knowledge and use of the Portfolio Diet and Portfolio Diet mobile application in clinical practice. Demonstrating that HCP rate the Portfolio Diet app as usable, educational, high quality, and has potential use in practice will further support clinical translation of the Portfolio Diet. This toolkit will also be used in the CIHR-funded Coronary Heart Effectiveness Assessment of the Portfolio diet in primary care (CHEAP) trial.

ELIGIBILITY:
Inclusion Criteria:

- Eligible participants are healthcare professionals that are registered with a regulatory college, including physicians, RDs, pharmacists and nurses.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-07-10 (Actual); Primary Completion 2024-08-12 (Actual); Study Completion 2024-08-12 (Actual)

PRIMARY OUTCOMES:
Face Validation | 30 minutes
  Face validity will be determined if <30% of respondents rating questions in parts B or C as either 1 or 2 (out of 5).
Content Validation | 30 minutes
  Content validity will be determined if <30% of respondents rating questions in part A of the phase 1 questionnaire as irrelevant.
Usability using the System Usability Scale | 8 days
  Usability will be determined using the System Usability Scale which ranges from 0 to 100 based on responses to 10 questions. An average System Usability Scale score of >70 indicates the tool being assessed is considered usable.
Usability using the mHealth App Usability Questionnaire | 8 days
  Usability will be determined using the standalone, HCP-facing MAUQ which includes 18 statements rated on a 7-point Likert scale. The total score will be calculated and an average score of the responses to all statements will be determined, with higher average scores indicating higher app usability.
Quality using the Mobile Application Rating Scale | 8 days
  Quality of the Portfolio Diet app will be determined using the Mobile Application Rating Scale (MARS) which comprises a 19-item objective evaluation across four domains: engagement, functionality, aesthetics, and information. The MARS also includes a 4-item subjective quality assessment, and a specific 6-item section tailored to the app being evaluated, all of which are rated on a 5-point Likert scale specific to each statement.
Knowledge Acquisition about the Portfolio Diet | 8 days
  A composite of 4 multiple-choice questions will be used to assess knowledge acquisition.
Engagement with the Portfolio Diet App | 8 days
  A composite of 11 open-ended and likert scale questions will be used to assess engagement with the app.
Acceptability of the Portfolio Diet App | 8 days
  A composite of 4 multiple-choice and open-ended questions will be used to assess acceptability of the portfolio diet and the app in specific patient populations.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Chiavaroli, PhD, Principal Investigator — University of Toronto
Locations (1):
- University of Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
To assess diversity and representation of marginalized groups serviced by our sample, we will include questions on whether HCP service these communities. We will also collect some information on the HCP to describe our sample, including age, sex, gender, ethnicity and type of HCP; however, we will use ranges or groupings of options as selections for responses to reduce identifiable information. No other personal information is collected. These data will be presented descriptively in the publication of results.

REFERENCES:
- [Background] Kavanagh ME, Chiavaroli L, Glenn AJ, Heijmans G, Grant SM, Chow CM, Josse RG, Malik VS, Watson W, Lofters A, Holmes C, Rackal J, Srichaikul K, Sherifali D, Snelgrove-Clarke E, Udell JA, Juni P, Booth GL, Farkouh ME, Leiter LA, Kendall CWC, Jenkins DJA, Sievenpiper JL. A Web-Based Health Application to Translate Nutrition Therapy for Cardiovascular Risk Reduction in Primary Care (PortfolioDiet.app): Quality Improvement and Usability Testing Study. JMIR Hum Factors. 2022 Apr 21;9(2):e34704. doi: 10.2196/34704. PMID 35451981
- [Background] Lynn MR. Determination and quantification of content validity. Nurs Res. 1986 Nov-Dec;35(6):382-5. No abstract available. PMID 3640358
- [Background] Chiavaroli L, Nishi SK, Khan TA, Braunstein CR, Glenn AJ, Mejia SB, Rahelic D, Kahleova H, Salas-Salvado J, Jenkins DJA, Kendall CWC, Sievenpiper JL. Portfolio Dietary Pattern and Cardiovascular Disease: A Systematic Review and Meta-analysis of Controlled Trials. Prog Cardiovasc Dis. 2018 May-Jun;61(1):43-53. doi: 10.1016/j.pcad.2018.05.004. Epub 2018 May 26. PMID 29807048
- [Background] Jenkins DJ, Kendall CW, Marchie A, Faulkner DA, Wong JM, de Souza R, Emam A, Parker TL, Vidgen E, Lapsley KG, Trautwein EA, Josse RG, Leiter LA, Connelly PW. Effects of a dietary portfolio of cholesterol-lowering foods vs lovastatin on serum lipids and C-reactive protein. JAMA. 2003 Jul 23;290(4):502-10. doi: 10.1001/jama.290.4.502. PMID 12876093
- [Background] Glenn AJ, Li J, Lo K, Jenkins DJA, Boucher BA, Hanley AJ, Kendall CWC, Shadyab AH, Tinker LF, Chessler SD, Howard BV, Liu S, Sievenpiper JL. The Portfolio Diet and Incident Type 2 Diabetes: Findings From the Women's Health Initiative Prospective Cohort Study. Diabetes Care. 2023 Jan 1;46(1):28-37. doi: 10.2337/dc22-1029. PMID 36162007
- [Background] Glenn AJ, Lo K, Jenkins DJA, Boucher BA, Hanley AJ, Kendall CWC, Manson JE, Vitolins MZ, Snetselaar LG, Liu S, Sievenpiper JL. Relationship Between a Plant-Based Dietary Portfolio and Risk of Cardiovascular Disease: Findings From the Women's Health Initiative Prospective Cohort Study. J Am Heart Assoc. 2021 Aug 17;10(16):e021515. doi: 10.1161/JAHA.121.021515. Epub 2021 Aug 4. PMID 34346245
- [Background] Pearson GJ, Thanassoulis G, Anderson TJ, Barry AR, Couture P, Dayan N, Francis GA, Genest J, Gregoire J, Grover SA, Gupta M, Hegele RA, Lau D, Leiter LA, Leung AA, Lonn E, Mancini GBJ, Manjoo P, McPherson R, Ngui D, Piche ME, Poirier P, Sievenpiper J, Stone J, Ward R, Wray W. 2021 Canadian Cardiovascular Society Guidelines for the Management of Dyslipidemia for the Prevention of Cardiovascular Disease in Adults. Can J Cardiol. 2021 Aug;37(8):1129-1150. doi: 10.1016/j.cjca.2021.03.016. Epub 2021 Mar 26. PMID 33781847
- [Derived] Viscardi G, Eskandari S, Chen A, Chiang N, Kavanagh ME, Back S, Vallis M, Scourboutakos MJ, Malik VS, Kendall CWC, Jenkins DJA, Sievenpiper JL, Chiavaroli L. Translating Cardiovascular Clinical Practice Guidelines on Nutrition Therapy: Validation of the Portfolio Diet Toolkit for Healthcare Providers. CJC Open. 2025 Sep 2;7(12):1662-1671. doi: 10.1016/j.cjco.2025.08.015. eCollection 2025 Dec. PMID 41542125